CLINICAL TRIAL: NCT06894992
Title: A Comparison of The Effectiveness of Tegoprazan and Lansoprazole in Achieving Cure Rates in Patients With Bleeding Peptic Ulcers: A Double-Blind Randomized Trial
Brief Title: Tegoprazan And Lansoprazole Effectiveness in Bleeding Peptic Ulcer Treatment
Acronym: TALENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Steffanus (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Sponsor-Investigator, Mario Steffanus, Gastroenterology and Hepatology Division Trainee, Dr Cipto Mangunkusumo General Hospital
Organization: Dr Cipto Mangunkusumo General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-12-1819
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Peptic Ulcer Bleeding
Keywords: Tegoprazan; Lansoprazole; Peptic Ulcer; Peptic Ulcer Bleeding; Healing Rate
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Peptic Ulcer | interventions — tegoprazan; Lansoprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potassium Channel Acid Blocker (Experimental): Each randomized patients will consume Tegoprazan 50 mg tab PO OD for 2 weeks
  Interventions: Drug: Tegoprazan
- Proton Pump Inhibitor (Active Comparator): Each randomized patients will consume Lansoprazole 30 mg tab PO OD for 2 weeks
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Tegoprazan — Tegoprazan 50 mg tab PO OD in 2 weeks
  Other Names: Potassium Channel Acid Blocker; PCAB
  Arms: Potassium Channel Acid Blocker
Drug: Lansoprazole — Lansoprazole 30 mg tab PO OD in 2 weeks
  Other Names: Proton Pump Inhibitor; PPI
  Arms: Proton Pump Inhibitor

SUMMARY:
The goal of this clinical trial is to compare the effects of tegoprazan vs lansoprazole in healing bleeding peptic ulcers. It will also teach about the safety of both modalities. The main questions it aims to answer are:

How does the effectiveness of Tegoprazan compare with Lansoprazole in two weeks of healing rate bleeding peptic ulcer patients in the Indonesian population?

Researchers will compare the drug tegoprazan to lansoprazole with a double-blind randomized control to see their effect on healing bleeding peptic ulcers.

Participants will:

Take drug tegoprazan 50 mg OD or lansoprazole 30 mg OD every day for 2 weeks Endoscopic examination at the beginning before treatment and after completion of treatment within 2 weeks Record of their adverse effect occurrence

DETAILED DESCRIPTION:
Peptic ulcer disease (PUD) is a condition characterized by disruption of the gastric and duodenal mucosal lining due to exposure to gastric acid or pepsin. Major causes include Helicobacter pylori infection, nonsteroidal anti-inflammatory drug (NSAID) use, gastric bypass surgery, lifestyle factors such as smoking and alcohol consumption, and genetic predisposition. PUD affects 5-10% of the global population and poses a significant healthcare burden, with prevalence rising from 6.43 million to 8.09 million cases between 1990 and 2019.

Current PUD treatment involves acid-suppressing agents and H. pylori eradication when indicated. Proton pump inhibitors (PPIs) play a key role by irreversibly inhibiting H⁺/K⁺ ATPase in gastric parietal cells, effectively maintaining gastric pH ≥4, which is essential for ulcer healing and preventing complications like bleeding. Lansoprazole, a widely used PPI, has demonstrated strong efficacy, with healing rates of 64%, 75.6%, and 95.7% at 2, 4, and 8 weeks, respectively. However, PPIs have limitations, including short plasma half-life, food dependency, breakthrough symptoms, and potential long-term adverse effects such as hypergastrinemia, acid rebound, and gut microbiota alterations.

To overcome these limitations, potassium-competitive acid blockers (PCABs) like vonoprazan and tegoprazan have been developed. PCABs provide faster, more stable, and potent acid suppression compared to PPIs. Unlike PPIs, which require activation in an acidic environment, PCABs directly inhibit H⁺/K⁺ ATPase by competitively binding to potassium sites, offering more predictable pharmacokinetics. Tegoprazan, a newer PCAB, has demonstrated superior acid suppression and a faster onset of action than vonoprazan, making it highly relevant for ulcer healing and preventing nocturnal acid breakthrough.

Studies suggest that PCABs are non-inferior to PPIs in treating PUD, with some data indicating that tegoprazan offers stronger, faster, and more stable acid suppression than vonoprazan. However, no studies have compared the healing rates of tegoprazan and lansoprazole specifically in bleeding PUD patients over a 2-week treatment period. Given the importance of optimizing treatment for bleeding PUD in Indonesia, this study aims to compare the effectiveness of tegoprazan and lansoprazole in ulcer healing over a short-term evaluation period.

This research is expected to contribute to the scientific literature by providing clinical trial data specific to the Indonesian population, inform clinical decision-making by identifying the most effective treatment for bleeding PUD, and ultimately improve patient outcomes by ensuring faster healing and better symptom management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with upper gastrointestinal bleeding caused by peptic ulcer through gastroscopic examination

Exclusion Criteria:

* Allergic to Tegoprazan or Lansoprazole
* Diagnosed with gastric or duodenal cancer, pregnant
* History of H. pylori infection treatment failure
* Presence of comorbidities such as chronic kidney disease or decompensated liver cirrhosis
* Alcohol consumption
* Undergoing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Healing Rate | 2 weeks
  The healing rate will be rated using Forrest Classification

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo National General Hospital, Jakarta, DKI Jakarta
  - Atma Jaya Hospital, Jakarta, DKI Jakarta

IPD SHARING:
Plan to Share IPD: Undecided